CLINICAL TRIAL: NCT04853719
Title: A Prospective, Randomized, Open-label, Multicenter Study Comparing Rivaroxaban 2.5 mg Twice Daily Associated With Aspirin 100 mg Once Daily Versus Aspirin 100 mg Once Daily in Patients With Peripheral Arterial Disease and Limiting Intermittent Claudication. (The COMPASS CLAUDICATION Trial).
Brief Title: Rivaroxaban 2.5 mg BID and Aspirin for Intermittent Claudication in PAD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Science Valley Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ScienceValley
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Intervention Model Description: 2 arms, active comparator (vascular dose) versus aspirin alone
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vascular dose (Experimental): Rivaroxaban 2.5 mg BID and aspirin 100 mg OD for 6 months
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet
- Aspirin (Active Comparator): Aspirin 100 mg OD for 6 months
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — oral anticoagulants plus antiplatelet agent
  Other Names: Aspirin 100 Mg oral Tablet

SUMMARY:
This trial is evaluating if rivaroxaban 2.5 mg BID and aspirin 100 mg OD compared to aspirin alone improves on intermittent claudication distance in PAD patients.

DETAILED DESCRIPTION:
Background: The COMPASS trial demonstrated that in patients with peripheral arterial disease the combination of rivaroxaban and aspirin compared with aspirin reduces the risk of major adverse limb events, but it is not known whether this combination can also improve symptoms in patients with intermittent claudication. The primary objective of this study is to evaluate the effect of the combination on intermittent claudication distance.

Study design: Eighty-eight patients with intermittent claudication will be randomized to receive rivaroxaban 2,5 mg twice daily plus aspirin 100 mg once daily or aspirin 100 mg once daily for 24 weeks. The primary outcome is the change in claudication distance from baseline to 24 hours as measured by 6 minutes walking test and treadmill test. The main safety outcome is the incidence of major bleeding according to ISTH criteria.

Summary: The COMPASS CLAUDICATION trial will provide high-quality evidence regarding the effect of the combination of rivaroxaban and aspirin on claudication distance in patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic PAD who signed the informed consent form (ICF) with:

  1. Ankle-brachial index (ABI) < 0. 85 in at least one member, and
  2. ACD < 500 meters
  3. age > 18 years
  4. No history of lower-limbs arterial bypass surgery or angioplasties in the last year
  5. walking ability limited by the symptom of claudication and
  6. ability to complete a treadmill test

Exclusion Criteria:

1. high risk of bleeding

   - Evidence of a recent history of bleeding in the last three months, hemorrhagic diathesis in the last three months, changes in coagulation tests (INR> 1.5 or aPTT > 2), pulmonary bronchiectasis, active cancer, active gastroduodenal ulcer, use of dual antiplatelet therapy.
2. Recent hemorrhagic stroke (1 month) or any history of previous hemorrhagic or lacunar stroke, if detected by occasional prior tomography, which is not part of the study protocol.
3. severe heart failure (NYHA class III and VI)
4. advanced stable kidney disease (estimated creatinine clearance <15 ml per minute), defined as eTFG <15 mL/min by 1.73 m2 calculated by the abbreviated formula Diet Modification in Kidney Disease (MDRD).
5. the use of dual antiplatelet therapy, anticoagulation, or other antithrombotic therapy
6. Continuous use of pentoxifylline or cilostazol
7. Cardiac conditions that may lead to heart failure, such as unstable angina, arrhythmias, acute myocardial infarction in the last three months
8. Non-cardiac conditions that may interfere with the ability to complete functional tests (e.g., chronic obstructive pulmonary disease, anemia, rheumatologic diseases)
9. Non-cardiovascular conditions are considered by the researcher as associated with a poor prognosis.

a. Active cancer with a life expectancy of fewer than six months b. Collagen limiting diseases c. Previous or scheduled surgeries that prevent functional evaluation d. Orthopedic diseases that hinder functional evaluation (j) Pregnancy. Women with the potential to bear children should be under contraceptive strategies and take a negative pregnancy test to be enrolled.

(k) Patients with COVID in the contagious phase (PCR+)

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total walking distance (TWD) at week 24 in meters in the 6-Minute Walk Test (6MWT) | 6 months

SECONDARY OUTCOMES:
Change from baseline in the total walking distance (TWD) at week 24 in meters in the treadmill test (TMT) | 6 months
Change from baseline in the Quality of Life Walking Impairment Questionnaire (WIQ) from at week 24 | 6 months

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE) | 6 months
  Exploratory Efficacy Outcome
Major Adverse Limb Events (MALE) | 6 months
  Exploratory Efficacy Outcome
Major or clinically non-relevant bleeding defined according to the International Society of Thrombosis and Hemostasis (ISTH) criteria | 6 months
  Primary Safety Outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital e Maternidade Christovão da Gama - Science Valley clinical site, Santo André, São Paulo
  - Science Valley Research Institute, Santo André, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All data is collected on RedCap, thast allows open and sharing IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year

REFERENCES:
- [Background] Ramacciotti E, Agati LB, Volpiani GG, Brito KF, Ribeiro CM, Aguiar VCR, Ramacciotti LS, Paganotti A, Pereira FM, Caffaro RA, Fioranelli A, Krakauer R, Rached HRS, Wolosker N, Anand SS, Eikelboom JW, Lopes RD. Rivaroxaban with Aspirin Versus Aspirin for Peripheral Arterial Disease and Intermittent Claudication. Rationale and Design of the COMPASS CLAUDICATION Trial. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296211073922. doi: 10.1177/10760296211073922. PMID 35043716
- [Derived] Ramacciotti E, Volpiani GG, Britto KF, Agati LB, Ribeiro CM, Aguiar VCR, Paganotti A, Pereira FM, Caffaro RA, Krakauer R, Rached HRS, Fareed J, Wolosker N, Anand SS, Eikelboom JW, Chang C, Lopes RD. Rivaroxaban for Patients with Intermittent Claudication. NEJM Evid. 2024 Sep;3(9):EVIDoa2400021. doi: 10.1056/EVIDoa2400021. Epub 2024 Aug 26. PMID 39185955